CLINICAL TRIAL: NCT02901106
Title: Monitoring of Patients Followed for a Multiple Sclerosis and Treated by Dimethyl-fumarate SURV-SEP
Brief Title: Monitoring of Patients Followed for a Multiple Sclerosis and Treated by Dimethyl-fumarate
Acronym: SURV-SEP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Another surveillance protocol was initiated by the OFSEP (OFSEP cohort) which allows to follow all the patients, whatever their treatment.
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JAB_2016_17
Record Dates: First submitted 2016-09-07; First posted 2016-09-15 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis, Relapsing-Remitting; Dimethyl fumarate
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with recurring-remitting MS (Experimental)
  Interventions: Drug: Dimethyl fumarate

INTERVENTIONS:
Drug: Dimethyl fumarate — Patient follow-up at 6, 12, 18, 36, and 60 months after the start of Dimethyl fumarate
  Systematization of cerebral MRI examination at 18 month and 5 years from the beginning of treatment by Dimethyl fumarate

SUMMARY:
The dimethyl fumarate is an oral drug, indicated in the treatment of the relapsing-remitting multiple sclerosis (MS) , which efficacy and safety has been assessed and validated in two randomised, placebo phase-controlled III international studies, organized by the pharmaceutical company developing the molecule. TECFIDERA® (dimethyl-fumarate) has received European approval on January 30, 2014, for the treatment of adult patients with relapsing remitting MS.

Treatment with dimethyl fumarate is introduced as part of the usual care under supervision of a physician experienced in the treatment of the disease.

It has proved effective to reduce the number of relapses in patients with recurring-remitting MS and reduce the number of patients who have relapses during treatment.

The objective of the study is to observe, in real conditions, on the one hand the tolerance and the other evolution, clinical and radiologic disease in patients already treated by dimethyl-fumarate and collect long-term safety data.

ELIGIBILITY:
Inclusion Criteria:

* patient 18 years old and more
* with multiple sclerosis according to the criteria of Mac Donald 2010 : relapsing-remitting (RR), secondary-progressive (SP) or primary-progressive (PP)
* for which treatment with dimethyl-fumarate has been prescribed
* followed at the Rothschild Foundation in the Neurology Department
* having given written consent to participation in the study

Exclusion Criteria:

* pregnant or breastfeeding woman
* patient with a measure of legal protection
* subject unaffiliated insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Number of patients with a relapse and/or progressive worsening of disease (EDSS score) | After one year of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmique Adolphe de Rothschild, Paris, France